CLINICAL TRIAL: NCT05580172
Title: A Phase 1 Open Label Dose Ranging Study of Oral RH324 in Advanced Non-Small Cell Lung Cancer
Brief Title: Phase 1 Study of Oral RH324 in Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ReHeva Biosciences,Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RHV18002
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): RH324
  Interventions: Drug: RH324
- Dose Level 2 (Experimental): RH324
  Interventions: Drug: RH324
- Dose Level 3 (Experimental): RH324
  Interventions: Drug: RH324

INTERVENTIONS:
Drug: RH324 — polymolecular

SUMMARY:
Phase 1 open label dose ranging study of RH324 in advanced non-small cell lung cancer

DETAILED DESCRIPTION:
This is a Phase 1 open label dose ranging study to assess the safety and tolerability of oral RH324 in advanced non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Advanced Non-Small Cell Lung Cancer
* Measurable Target Lesion by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Failed all standard of care including chemotherapy, targeted therapy, and immunotherapy
* Adults over 18 years
* Performance status (Eastern Cooperative Oncology Group) less than or equal to 2
* Life expectancy greater than 2 months
* Laboratory Values:

Hemoglobin greater than or equal to 9; neutrophils greater than 1,000; platelets greater than 50,000 Liver function tests less than or equal to twice upper limit of normal Serum Creatinine less than or equal to 2 Creatinine clearance greater than or equal to 30 mL per minute Hemoglobin A1C less than 7 Normal Thyroid function

* No history of hyperthyroidism
* Abstinence from alcohol and supplements
* Not pregnant, lactating and willing to use birth control throughout study
* Able to provide consent
* Positive Emission Tomography/Computer Tomography part of subjects care plan at baseline

Exclusion Criteria:

* Prior use of Withania somnifera
* Phenylketonuria
* Inability to swallow capsules
* Hypersensitivity to study drug ingredients
* Unstable medical or surgical condition
* History of additional cardiac risk factors
* Requiring drugs that are "strong" inhibitors of cytochrome P450
* Requiring irradiation
* Requiring intravenous fluids or hyperalimentation
* Requiring transfusions, dialysis, or other procedures
* Active infection
* Human Immunodeficiency Virus
* Must exceed washout period of prior treatments
* Psychiatric, neurological or other reason that precludes subjects ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Per Common Terminology Criteria for Adverse Events Version 5 | Through Study Completion 28 Days
  Percentage of Adverse Events Summarized by Causality and Grade

SECONDARY OUTCOMES:
Percentage of Subjects with a Change from Baseline on Physical Examination and Vital Signs | Through Study Completion 28 Days
  Percentage of Subjects with a Clinically Relevant Change from Baseline on Physical Exam and Vital Signs
Percentage of Subjects with a Change from Baseline on Laboratory Values | Through Study Completion 28 Days
  Percentage of Subjects with a Clinically Relevant Change from Baseline on Blood and Urine Laboratory Values
Percentage of Subjects with a Change from Baseline on the Electrocardiogram | Through Study Completion 28 Days
  Percentage of Subjects with a Clinically Relevant Change from Baseline on the 12-Lead Electrocardiogram
Percentage of Subjects with a Change from Baseline in Quality of Life | Through Study Completion 28 Days
  Percentage of Subjects with a Clinically Relevant Change from Baseline in Quality of Life Based on the Eastern Cooperative Oncology Group Performance Status Levels

CONTACTS AND LOCATIONS:
Locations (1):
- Case Comprehensive Cancer Center University Hospitals, Cleveland, Ohio, United States